CLINICAL TRIAL: NCT04185207
Title: Study on the Relationship Between Chinese Women's Perinatal Mental Health and Socioeconomic Status
Acronym: ACWPMHSS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Collaborators: Gansu Provincial Maternal and Child Health Care Hospital (Other)
Responsible Party: Principal Investigator, Hongbo Qi, Director of Obstetric, First Affiliated Hospital of Chongqing Medical University
Other Study IDs: Q20191025
Record Dates: First submitted 2019-10-29; First posted 2019-12-04 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Mental Disorders During Pregnancy; Mental Disorder in the Puerperium - Baby Delivered
Keywords: Mental health; Socioeconomic status
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — There is no intervention.

SUMMARY:
The objective of this study is to explore the relationship between perinatal women's mental health and socioeconomic status, observe the perinal outcomes of different income level, and make mental health reference value for them. Questionaires will be used to investigate women's income and mental health status in 4 periods, including the first, second, third trimester and postpartum 42 days. After delivery, birth outcomes will be collected from participating hospitals' clinical case system. All data will be analysed with statistical software.

DETAILED DESCRIPTION:
The objective of this study is to explore the relationship between perinatal women's mental health and socioeconomic status, observe the perinal outcomes of different income level, and make mental health reference value for them. Several hospitals from 5 provinces located in the est, west, south, north and middle of China will participate in the study which plans to include 5000 pregnant women. Questionaire will be used to investigate women's income and mental health status in 4 periods, including the first, second, third trimester and postpartum 42 days. After delivery, birth outcomes will be collected from participating hospitals' clinical case system. All data will be analysed with statistical software.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to read and understand informed consent; Age 18-59; Singleton in 12-14 gestational weeks; Plan to give bith in participating hospital; Must be able to comply with study regulations;

Exclusion Criteria:

* Unmarried women; Multiple-pregnancy; Clinical diagnosis of mental disorders before;

Ages: 18 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant women;
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Income level of perinatal women | 1 year
  A questionnaire investigation on the income in 5 participating hospitals will be conducted. The minimum value is 0 and the maximum value is over than 10000 RMB. It is used to investigate income level.

SECONDARY OUTCOMES:
Pregnancy stress | 1 year
  This will be measured with Pregnancy Stress Rating Scale. The response options for each item indicate the level of prenatal stress ranging from 0-no stress to 3-severe stress. The results are the average score of all items, and higher scores indicate the higher level, with 0 for no stress, 0.01-1.00 for mild stress, 1.01-2.00 for moderate stress and 2.01-3.00 for severe stress.
Pregnancy anxiety | 1 year
  This will be measured with the scale of Generalized Anxiety Disorder-7, GAD-7. GAD-7 consisted of seven questions where each question is rated on a scale (0 - 3), three being the maximum. Each subject had a total summed score across all the seven dimensions which range between 0 and 21, a higher score indicates a higher level of anxiety, with 0-4 for no anxiety, 5-9 for mild anxiety, 10-14 for moderate anxiety and 15-21 for severe anxiety.
Pregnancy depression | 1 year
  This will be measured with the scale of Patient Health Questionnaire-9（PHQ-9）. There are 9 questions in the scale where each question is rated on a scale (0-3), with a high sensitivity and speciality while reaching a cutoff score of 10. Responses are summed to obtain a total score that can range from 0 to 27; scores of 5, 10, 15, and 20 serve as cutoff scores that indicate mild, moderate, moderately severe, and severe depression.
Pregnancy somatic symptoms | 1 year
  Screening for somatization disorders and assessing the severity of somatic symptoms with the scale of Patient Health Questionnaire-15（PHQ-15）. There are 15 items in the scale where each item is rated on a scale 0(none)-2(massive). Responses are summed to obtain a total score that range from 0 to 30, with 0-4 for no symptom, 5-9 for mild symptom, 10-14 for moderate symptom and 15-30 for severe symptom.
Quality of life in pregnancy | 1 year
  Perinatal women's quality of life will be measured with the three-level version of European Quality of life five-dimensional scale(EQ-5D-3L). Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jianlin ZHAO, Study Director — First Affiliated Hospital of Chongqing Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mei-Dan E, Ray JG, Vigod SN. Perinatal outcomes among women with bipolar disorder: a population-based cohort study. Am J Obstet Gynecol. 2015 Mar;212(3):367.e1-8. doi: 10.1016/j.ajog.2014.10.020. Epub 2014 Oct 15. PMID 25446660
- [Result] Glover V, O'Donnell KJ, O'Connor TG, Fisher J. Prenatal maternal stress, fetal programming, and mechanisms underlying later psychopathology-A global perspective. Dev Psychopathol. 2018 Aug;30(3):843-854. doi: 10.1017/S095457941800038X. PMID 30068411
- [Result] Rocheleau CM, Bertke SJ, Lawson CC, Romitti PA, Desrosiers TA, Agopian AJ, Bell E, Gilboa SM; National Birth Defects Prevention Study. Factors associated with employment status before and during pregnancy: Implications for studies of pregnancy outcomes. Am J Ind Med. 2017 Apr;60(4):329-341. doi: 10.1002/ajim.22700. PMID 28299820